CLINICAL TRIAL: NCT06290921
Title: Ovulation Trigger With Less Than 3 Follicles in Stimulated In-vitro Fertilization (IVF) Cycles
Brief Title: Ovulation Triggering 2 vs 3 Follicles
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3472
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ovulation triggering — Ovulation triggering when women only 2 dominant follicles as opposed to the clinic's standard of 3 follicles or more

SUMMARY:
Poor responders in in-vitro fertilization (IVF) cycles represent a major challenge for fertility specialists. Although poor responders tend to have sub-optimal fertility treatment outcomes, many of these patients wish to attempt at least one IVF cycle. Traditionally, IVF cycles producing less than 3 to 4 mature follicles (measuring at least 14 mm) have either been cancelled or converted to intra-uterine insemination (IUI) due to the low pregnancy rates associated with these cycles. The minimal number of follicles required to proceed with egg collection is based on clinical experience, having been determined by weighing the probability of implantation and pregnancy versus the risk of not obtaining quality oocytes or reaching embryo transfer when fewer mature follicles are present. This retrospective quality control study aims to compare pregnancy rates in IVF cycles producing 3 follicles measuring 14 mm and more on trigger day, versus 2 or fewer follicles.

ELIGIBILITY:
Inclusion Criteria:

* Stimulated IVF cycle at clinique ovo
* Patients with a maximum of 3 mature follicles (≥14mm) on the day of ovulation trigger

Exclusion Criteria:

* Cycle cancelation due to no follicles
* History of recurrent implantation failure
* Contraindication of ovulation induction medication

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women able to have an embryo transfered in their uterus
Study Population: Data spreadsheet from 2011 to 2017 of patients having undergone an IVF cycle
Sampling Method: Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 6 to 8 weeks after Frozen Embryo Transfer
  clinical pregnancy is the presence of fetal heartbeat at the viability ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Louise Lapensée, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No